CLINICAL TRIAL: NCT01006330
Title: Dysphagia in Elderly Medical Patients: Occupational Therapy Evaluation and Prevalence
Brief Title: Dysphagia in Elderly Medical Patients
Acronym: DEM
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Tina Hansen, MSc.OT, Herlev Hospital
Other Study IDs: CVR29190623; HC-2009-061 (Registry Identifier: The local ethical committee in the Capital region)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2009-10

CONDITIONS: Deglutition Disorders; Impaired Cognition; Physical Activity; Complete Immobility Due to Frailty; Respiratory Tract Infections
MeSH Terms: conditions — Deglutition Disorders; Cognition Disorders; Motor Activity; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elderly medical inpatients

SUMMARY:
Dysphagia in hospitalized elders is associated with less positive outcomes in rehabilitation, increased likelihood of readmission, increased comorbidity and mortality, and increased length of hospital stay. In light of an increase in the elderly population in Denmark, the consequences of dysphagia, and the importance of minimizing the risk of disability and frailty, it is vital to emphasize safe participation of the elderly dysphagic patient in eating, drinking and swallowing. Danish occupational therapists have an important role in the dysphagia management, but no Danish evidence-based occupational therapy assessments for dysphagia of elderly medical patients exist. In order to oblige this lack, the objective of the study is to provide an assessment tool with operational definitions of dysphagia which includes the complexity of performance in eating, drinking and swallowing, is evidence-based, and guides occupational therapists in the treatment planning in a client-centred and purposeful manner.

The study involves a quantitative approach, and is initiated by a translation and cultural adaptation of the Canadian "The McGill Ingestive Skills Assessment" (MISA). Hereafter, the psychometric qualities are tested. On basis of the data collected for the psychometrics, the prevalence and characteristics of dysphagia in the study population are investigated. Provided that the psychometric testing of the MISA reveals satisfactory levels, the effect of using the MISA in the treatment planning is investigated.

It is hypothesized that:

The Danish translation of the MISA will demonstrates satisfactory content validity, reliabilities, convergent validity, known-groups validity, predictive validity, criterion validity, high levels of sensitivity/specificity and are responsive to change.

Dysphagia is prevalent in elderly medical patients at the time of admission to acute medical care and there can be found a correlation between dysphagia severity and the presence of comorbidity, disability, frailty, the length of hospital stay, the place of discharge and the number of readmissions for elderly medical patients.

DETAILED DESCRIPTION:
The study is divided into four study parts.

Study I aims to translate and cultural adapt the MISA into Danish occupational therapy terminology, to secure equivalency between the original and the translated version, and to test its interrater- and intrarater reliability as well as internal consistency.

Study II aims to investigate the convergent validity, known-groups validity, predictive validity and the responsiveness of the MISA.

Study III aims to test the criterion-related validity and the diagnostic accuracy of the MISA using the Flexible Endoscopic Evaluation of Swallowing (FEES) and the Assessment of Motor and Process Skills (AMPS) as gold standards; and to compare the diagnostic accuracy for aspiration of the MISA compared to the Water Swallow Test, when using the FEES as the gold standard.

Study IV aims to investigate the prevalence and characteristics of dysphagia in elderly medical patients, and to identify its potential associations between comorbidity, disability, frailty, length of hospital stay, place of discharge and number of readmissions.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years
* needs > 2 days of hospitalization
* are able to give personal information regarding self, place and time
* are alert > 30 minutes
* are able to maintain an upright seating position and head control
* are able to swallow saliva spontaneously and on command
* are able to voluntary cough or clear the throat twice
* working knowledge of the Danish language
* consent to participate and able to give written informed consent.

Exclusion criteria:

* needs oral/pharyngeal suctioning
* use of tube feeding for more than half of the caloric requirements
* tracheostomy
* terminally ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 102 internal medical patients admitted to Herlev Hospital are included consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hansen, MSc PHD stud, Principal Investigator — Herlev Hospital, Region H
Locations (1):
- Occupational Therapy department, Herlev Hospital, Herlev, The Capital Region, Denmark